CLINICAL TRIAL: NCT02447822
Title: A Prospective Randomized Controlled Study to Evaluate Feasibility and Safety of Early Steroid Withdrawal After 6mg/kg vs 4.5mg/kg Thymoglobulin Induction Therapy in Kidney Transplantation
Brief Title: Thymoglobulin Induction Therapy in Kidney Transplantation (6mg/kg vs 4mg/kg)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Duck Jong Han, Professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AsanMC 2014-1213
Record Dates: First submitted 2015-05-15; First posted 2015-05-19 (Estimated); Last update posted 2015-05-19 (Estimated); Status verified 2015-05

CONDITIONS: Kidney Failure
MeSH Terms: conditions — Renal Insufficiency | interventions — thymoglobulin

ARMS (2):
- 6.0ATG (Active Comparator): Recipients who have 6.0 mg/kg Thymoglobulin as induction therapy
  Interventions: Drug: Thymoglobulin
- 4.5ATG (Active Comparator): Recipients who have 4.5 mg/kg Thymoglobulin as induction therapy
  Interventions: Drug: Thymoglobulin

INTERVENTIONS:
Drug: Thymoglobulin — 6.0 mg/kg vs 4.5 mg/kg Thymoglobulin

SUMMARY:
This is a prospective randomized controlled study to evaluate feasibility and safety of early steroid withdrawal after 6mg/kg vs 4.5mg/kg Thymoglobulin induction therapy in kidney transplantation. Patients are enrolled from June, 2015 for 24 months. They are randomized to either 6mg/kg or 4.5mg/kg Thymoglobulin induction group. Steroid withdrawal is done within one week after kidney transplantation for all the patients. Maintenance immunosuppressants are Tacrolimus and Mycophenolate mofetil (or Myfortic). Primary outcome is a composite of biopsy-proven acute rejection, delayed graft function, graft loss or death within one year post transplant.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients with renal failure from 18 to 70 years of age
* Candidates for cadaveric or living donor kidney transplantation
* Patients who are able and willing to consent the protocol of the study

Exclusion Criteria:

* Patients who have been receiving immunosuppressive therapy before transplantation
* Patients who have received an investigational medication within the past 30 days
* Patients who have a known contraindication to the administration of antithymocyte globulin
* Patients who are suspected or known to have an infection or were seropositive for hepatitis B surface antigen (HBsAg), antibody against hepatitis B core antigen (anti-HBcAg), hepatitis C virus (HCV), or human immunodeficiency virus (HIV)
* Patients who have had cancer (except non melanoma skin cancer) within the previous 2 years
* Pregnant women, nursing mothers, and women of childbearing potential who were not using condoms or oral contraceptives

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2015-06; Primary Completion 2018-05 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
A composite outcome of biopsy-proven acute rejection, delayed graft function, graft loss, and death | 12 months after kidney transplantation

SECONDARY OUTCOMES:
Pathologic findings according to Banff 2013 criteria | 1 day at the time of biopsy
Overall rate of acute rejection | 12 months after kidney transplantation
The rate of steroid-free immunosuppressive regimen | 12 months after kidney transplantation

REFERENCES:
- [Derived] Ko Y, Wee YM, Shin S, Kim MJ, Choi MY, Kim DH, Lim SJ, Jung JH, Kwon H, Kim YH, Han DJ. A prospective, randomized, non-blinded, non-inferiority pilot study to assess the effect of low-dose anti-thymocyte globulin with low-dose tacrolimus and early steroid withdrawal on clinical outcomes in non-sensitized living-donor kidney recipients. PLoS One. 2023 Mar 1;18(3):e0280924. doi: 10.1371/journal.pone.0280924. eCollection 2023. PMID 36857393